CLINICAL TRIAL: NCT00510666
Title: Butorphanol and Tramadol for Morphine PCA Pain Management After Total Hysterectomy
Brief Title: Comparison of Butorphanol and Tramadol Associated Patient-Controlled Analgesia (PCA) After Hysterectomy
Acronym: BATPCAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-2579-3FW; NMU2007092
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Postoperative Pain; Hysterectomy
Keywords: Pain, Postoperative; Analgesics, Opioid; Analgesia, Patient-Controlled; Pain Measurement
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Sodium Chloride; Butorphanol; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Butorphanol basal infusion adjunct to morphine PCA
  Interventions: Drug: Butorphanol tartrate
- 2 (Experimental): Saline infusion adjunct to morphine PCA
  Interventions: Drug: Saline
- 3 (Experimental): Premedication of Tramadol
  Interventions: Drug: Tramadol Hydrochloride
- 4 (Experimental): Preemptive saline for morphine PCA
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — Saline infusion adjunct to morphine PCA pump
  Other Names: SA
  Arms: 2
Drug: Butorphanol tartrate — Butorphanol was delivered at a continuous infusion manner adjunct to morphine PCA pump
  Other Names: BT
  Arms: 1
Drug: Tramadol Hydrochloride — 100mg tramadol was used preemptively to morphine PCA pump
  Other Names: TH
  Arms: 3
Drug: Saline — Preemptive saline as a control group to tramadol one
  Other Names: PS
  Arms: 4

SUMMARY:
Intravenous patient-controlled analgesia (PCA) is a popular technique for postoperative pain management. Although several drugs are recognized as effective therapeutic options, optimal selection of drugs in hysterectomy patients underwent different anesthesia treatments remains unknown explicitly. The investigators hypothesized that butorphanol and tramadol can produce different analgesic effects with intravenous PCA after abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Chinese
* 19-64yr
* Uterus myoma

Exclusion Criteria:

* Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records.
* Participants younger than 18yr，older than 65yr or pregnancy was eliminated.
* Due to the significant changes in vital signs might affect cognition of pain and that of sensation, over 20% variation of these records from the baselines or below 92% of SpO2 under 20-40% nasal tube oxygen at any time should be excluded from the study.
* Those who were not willing to or could not finish the whole study at any time.
* Any patient who exhibited a combative or incoherent state of PCA analgesia would be excluded from the study.
* Allergy to local anesthetics.
* Failed to perform the epidural catheterization.
* Those who demonstrated significant nerve-associated side effects from the insertion of the epidural needle.

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 841 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
VAS pain scoring; | 5 months

SECONDARY OUTCOMES:
VAS sedation scoring; VAS happiness scoring; Adverse effects; Patient's overall conditions. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Wang F, Shen X, Liu Y, Xu S, Guo X. Continuous infusion of butorphanol combined with intravenous morphine patient-controlled analgesia after total abdominal hysterectomy: a randomized, double-blind controlled trial. Eur J Anaesthesiol. 2009 Jan;26(1):28-34. doi: 10.1097/EJA.0b013e32831a6aa2. PMID 19122548